CLINICAL TRIAL: NCT02575404
Title: Phase IB Study of a Galectin Inhibitor (GR-MD-02) and Pembrolizumab in Patients With Metastatic Melanoma, Non-Small Cell Lung Cancer, and Head and Neck Squamous Cell Carcinoma.
Brief Title: GR-MD-02 Plus Pembrolizumab in Melanoma, Non-small Cell Lung Cancer, and Squamous Cell Head and Neck Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Galectin Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-166
Record Dates: First submitted 2015-10-09; First posted 2015-10-14 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Melanoma; Non-Small Cell Lung Cancer; Squamous Cell Carcinoma of the Head and Neck
Keywords: Metastatic; Keytruda; pembrolizumab; GR-MD-02; Galactoarabino-rhamnogalacturonate; Immunotherapy
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis | interventions — belapectin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2 mg/kg GR-MD-02 (Experimental): 2 mg/kg GR-MD-02 in combination with standard pembrolizumab treatment.
  Interventions: Drug: GR-MD-02; Drug: Pembrolizumab
- 4 mg/kg GR-MD-02 (Experimental): 4 mg/kg GR-MD-02 in combination with standard pembrolizumab treatment.
  Interventions: Drug: GR-MD-02; Drug: Pembrolizumab
- 8 mg/kg GR-MD-02 (Experimental): 8 mg/kg GR-MD-02 in combination with standard pembrolizumab treatment.
  Interventions: Drug: GR-MD-02; Drug: Pembrolizumab
- 4 mg/kg GR-MD-02 17 Cycles Maximum (Experimental): 4 mg/kg GR-MD-02 in combination with standard pembrolizumab treatment up to a maximum of 17 cycles.
  Interventions: Drug: GR-MD-02; Drug: Pembrolizumab

INTERVENTIONS:
Drug: GR-MD-02 — Patients will receive five doses of GR-MD-02 intravenously over 85 Days.
  Other Names: Galactoarabino-rhamnogalactouronate
Drug: Pembrolizumab — Patients will receive five 200mg doses of pembrolizumab intravenously over 85 days. After 85 days, patients may continue to receive pembrolizumab every 3 weeks if clinical benefit is noted.
  Other Names: Keytruda

SUMMARY:
This study is a dose escalation of GR-MD-02 with the standard therapeutic dose of pembrolizumab in patients with advanced melanoma, non-small cell lung cancer, and head and neck squamous cell cancer.

DETAILED DESCRIPTION:
This study will employ a 3+3 phase I design with dose escalation of GR-MD-02 in conjunction with the standard therapeutic dose of pembrolizumab in patients with advanced melanoma who have had progression after ipilimumab and/or BRAF targeted therapy when a BRAF mutation is present, non-small cell lung cancer patients with disease progression after targeted therapy, or head and neck squamous cell carcinoma patients with disease progression after at least one platinum-containing regimen.

In addition to monitoring for toxicity and clinical response, blood and tumor samples will be obtained to assess immunologic measures relevant to galectin biology and pembrolizumab T-cell checkpoint inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic or unresectable melanoma for whom treatment with pembrolizumab is indicated. Histological confirmation of melanoma will be required by previous biopsy or cytology.
* Patients with non-small cell lung cancer for whom treatment with pembrolizumab is indicated.
* Patients with squamous cell carcinoma of the head and neck for whom treatment with pembrolizumab is indicated
* Patients who have radiographic progression using Response Evaluation Criteria In Solid Tumors (RECIST) currently on pembrolizumab are also eligible.
* Patients must be ≥ 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Women of childbearing potential must have a serum or urine pregnancy test performed within 72 hours prior to the start of protocol treatment. The results of this test must be negative in order for the patient to be eligible. In addition, women of childbearing potential as well as male patients must agree to take appropriate precautions to avoid pregnancy.
* No active bleeding.
* Anticipated lifespan greater than 12 weeks.
* Patients must sign a study-specific consent document.

Exclusion Criteria:

* Patients who have previously received a galectin antagonist
* Patients with active autoimmune disease except for autoimmune thyroiditis or vitiligo
* Patients with history of colitis
* Patients with untreated brain metastases. Patients with treated brain metastases who demonstrate control of brain metastases with follow-up imaging 4 or more weeks after initial therapy are eligible.
* Other active metastatic cancer requiring treatment.
* Patients with active infection requiring antibiotics.
* Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus.
* Need for chronic steroids. Inhaled corticosteroids are acceptable.
* Laboratory values (to be performed within 28 days of enrollment) outside of protocol-specified ranges.
* Inability to give informed consent and comply with the protocol. Patients with a history of psychiatric illness must be judged able to understand fully the investigational nature of the study and the risks associated with the therapy.
* Any medical condition that in the opinion of the Principal Investigator would compromise the safety or conduct of the study procedures.
* Unresolved immune-mediated pneumonitis, diarrhea, elevation of hepatocellular enzymes or other toxicities requiring greater than physiological replacement doses of steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Frequency and Severity of Treatment-Related Adverse Events Measured by Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 | 85 Days
  Patients are seen in clinic 7 times over 85 days. At each visit, a research nurse performs a toxicity check. Patients have 5 physical exams during the 85-day period.

SECONDARY OUTCOMES:
Measure the response rate to combined therapy with GR-MD-02 and pembrolizumab in patients. | Baseline and at Day 85
  Patients will have PET and CT scans at baseline and after 85 days to assess response to treatment.
Assess the biological activity of GR-MD-02 in combination with pembrolizumab. | 85 Days
  Patients will provide 5 blood samples over 85 days to measure the absolute number of CD4+T Cells, CD8+ T cells and melanoma-specific T cells

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Curti, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Cancer Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Providence Cancer Center — http://oregon.providence.org/our-services/p/providence-cancer-center/